CLINICAL TRIAL: NCT02442232
Title: Hemodynamic Changes After Anesthesia With Propofol: Study of Biomarkers
Status: Completed | Type: Observational
Sponsor: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Gustavo Henrique Oliveira de Paula, PhD student, University of Sao Paulo
Other Study IDs: CNPq
Record Dates: First submitted 2015-05-07; First posted 2015-05-13 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Hemodynamic Responses to Propofol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Normotensive
- Hypertensive taking ACEi
- Hypertensive not taking ACEi

SUMMARY:
The purpose of this study is to evaluate biomarkers affecting the hemodynamic responses to propofol. Particularly, the investigators will assess the effects of polymorphisms in NOS3 and PRKCA genes on hemodynamic responses to propofol and the effects of these polymorphisms on biomarkers related to nitric oxide after propofol anesthesia. In addition, the investigators will evaluate the effects of propofol anesthesia on biomarkers related to nitric oxide in hypertensive patients chronically treated with angiotensin-converting enzyme inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II
* BMI lower 30 kg/m2

Exclusion Criteria:

* Severe hypertension
* Previous stroke
* Previous infarction
* Uncontrolled respiratory, renal, hepatic and hematological diseases.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients under propofol anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | 10 minutes
Diastolic blood pressure | 10 minutes
Mean blood pressure | 10 minutes
Heart rate | 10 minutes
Plasma nitrite levels | 10 minutes
Plasma nitrate levels | 10 minutes

REFERENCES:
- [Derived] Oliveira-Paula GH, Coeli-Lacchini FB, Ferezin LP, Ferreira GC, Pinheiro LC, Paula-Garcia WN, Garcia LV, Tanus-Santos JE, Lacchini R. Arginase II polymorphisms modify the hypotensive responses to propofol by affecting nitric oxide bioavailability. Eur J Clin Pharmacol. 2021 Jun;77(6):869-877. doi: 10.1007/s00228-020-03059-9. Epub 2021 Jan 7. PMID 33410970